CLINICAL TRIAL: NCT06589063
Title: Transcatheter Aortic Valve Replacement in Severe Low Flow, Low Gradient Aortic Stenosis: the Multicenter LOW-TAVR Registry
Brief Title: Transcatheter Aortic Valve Replacement in Severe Low Flow, Low Gradient Aortic Stenosis
Acronym: LOW-TAVR
Status: Recruiting | Type: Observational
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Gennaro Galasso, Professor, University of Salerno
Other Study IDs: 13202409
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Low Flow, Low Gradient Aortic Stenosis
Keywords: aortic stenosis; transcatheter aortic valve replacement; clinical outcomes; interventional cardiology
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Transcatheter aortic valve replacement — Transcatheter aortic valve replacement with implantation of new-generation balloon-expandable or self-expandable bioprostheses
  Other Names: TAVI; TAVR; Transcatheter aortic valve implantation

SUMMARY:
LOW-TAVR is a real-world, retrospective and prospective, multicenter Italian registry aimed at evaluating the characteristics and clinical outcomes of patients with severe low flow, low gradient aortic stenosis undergoing transcatheter aortic valve replacement (TAVR) and, in particular:

* risk factors
* gender differences
* comorbidities
* pharmacological treatment
* TAVR procedural characteristics
* periprocedural and in-hospital complications
* clinical outcome at 30-day, 1-year, 2-year and 5-year follow-up

DETAILED DESCRIPTION:
LOW-TAVR is a real-world, retrospective and prospective, multicenter Italian registry aimed at evaluating the characteristics and clinical outcomes of patients with severe low flow, low gradient aortic stenosis (LFLG-AS) undergoing transcatheter aortic valve replacement (TAVR).

The register aims to include at least 1,500 patients diagnosed with LFLG-AS undergoing TAVR at the participating centres.

The inclusion criteria are:

* LFLG-AS diagnosis according to current European Society of Cardiology guidelines
* Age 18 years or older
* Written informed consent

The exclusion criteria are:

* LFLG-AS pseudo-severe or non-confirmed severe aortic stenosis
* LFLG-AS referred for medical treatment or undergoing surgery

Clinical outcome is evaluated at a 30-day, 1-year, 2-year, and 5-year follow-up.

The primary endpoint of interest of the registry is the assessment of the incidence of the composite of all-cause mortality and hospitalization for heart failure at one year.

The secondary endpoints are the assessment of:

* periprocedural TAVR complications: complete atrioventricular block, stroke, acute myocardial infarction, acute aortic insufficiency, cardiogenic shock, acute pulmonary edema, cardiac tamponade, aortic rupture;
* adverse events during hospitalization: major and minor bleeding, major and minor vascular complications, definitive pacemaker implantation, cardiogenic shock, myocardial infarction, stroke, and death;
* adverse events at 30 days, one year, two years, and five years: all-cause mortality, hospitalizations for heart failure, cardiovascular mortality, myocardial infarction, stroke, major and minor bleedings.

ELIGIBILITY:
Inclusion Criteria:

* LFLG-AS diagnosis according to current European Society of Cardiology guidelines
* Age 18 years or older
* Written informed consent

Exclusion Criteria:

* LFLG-AS pseudo-severe or non-confirmed severe aortic stenosis
* LFLG-AS referred for medical treatment or undergoing surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe low flow, low gradient aortic stenosis (LFLG-AS) undergoing transcatheter aortic valve replacement (TAVR)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause death and hospitalization for worsening heart failure | 1 year
  Death due to cardiac or non-cardiac cause and new hospitalization for worsening heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salerno, Salerno, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT06589063/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT06589063/ICF_001.pdf